CLINICAL TRIAL: NCT04102371
Title: Pragmatic Pediatric Trial of Balanced Versus Normal Saline Fluid in Sepsis
Acronym: PRoMPT BOLUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Boston Children's Hospital (Other); Children's Healthcare of Atlanta (Other); Children's Hospital Colorado (Other); Children's Hospital Los Angeles (Other); University of Pittsburgh (Other); Morgan Stanley Children's Hospital (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); Children's Medical Center Dallas (Other); Children's National Research Institute (Other); Children's Hospital Medical Center, Cincinnati (Other); Hasbro Children's Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Nationwide Children's Hospital (Other); Primary Children's Hospital (Other); Seattle Children's Hospital (Other); St. Louis Children's Hospital (Other); Baylor College of Medicine (Other); University of California, Davis (Other); University of California, San Francisco (Other); University of Michigan (Other); Kidz First Hospital Middlemore (Unknown); Gold Coast Hospital and Health Service (Other Government); Queensland Children's Hospital (Other Government); Westmead Children's Hospital (Unknown); Sydney Children's Hospitals Network (Other); Perth Children's Hospital (Unknown); Starship Children's Hospital (Unknown); Monash Children's Hospital (Unknown); Women's and Children's Hospital, Australia (Other Government); Royal Children's Hospital (Other); Royal Darwin Hospital (Unknown); M.D. Anderson Cancer Center (Other); Virginia Commonwealth University (Other); Alberta Children's Hospital (Other); British Columbia Children's Hospital (Other); Centre Hospitalier Univeritaire Sainte Justine (Unknown); Centre Hospitalier Universitaire de Quebec (Unknown); Children's Hospital of Eastern Ontario (Other); The Hospital for Sick Children (Other); IWK Health Centre (Other); Jim Pattison Children's Hospital (Unknown); Kingston Health Sciences Centre (Other); London Health Sciences Centre (Other); McMaster Children's Hospital (Other); Stollery Children's Hospital (Other); The Children's Hospital of Winnipeg (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Pennsylvania Department of Health (Other Government); Townsville University Hospital (Other)
Responsible Party: Principal Investigator, Frances Balamuth, Principal Investigator, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-016484; R01HD101528 (NIH)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Shock; Septic
Keywords: Sepsis; Septic Shock; Fluid resuscitation; Saline; Balanced Fluid; Mortality; Crystalloid; PlasmaLyte; Lactated Ringer's; Kidney injury
MeSH Terms: conditions — Shock; Sepsis; Shock, Septic | interventions — Ringer's Lactate; Saline Solution; Plasma-lyte 148

STUDY DESIGN:
Intervention Model Description: Multi-center, open-label, randomized pragmatic comparative effectiveness trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Balanced fluids (BF) (Experimental): Balanced fluids (BF), including Lactated Ringer's and Plasma-Lyte (PL), will be administered to patients randomized to the experimental arm. BF will be used for all fluid boluses and maintenance fluids (supplemental electrolytes are allowed) from time immediately after randomization through 11:59 pm of the next calendar day. The determination of when to give fluid, how much fluid to give, how fast to give fluid, and what access to use to administer fluid will remain at the discretion of the treating team.
  Interventions: Drug: Lactated Ringer; Drug: Plasma-lyte
- 0.9% "Normal" Saline Fluid (NS) (Active Comparator): 0.9% "normal" saline (NS) fluid will be administered to patients randomized to the active comparator (control) arm. NS will be used for all fluid boluses and maintenance fluids (supplemental electrolytes are allowed) from time immediately after randomization through 11:59 pm of the next calendar day. The determination of when to give fluid, how much fluid to give, how fast to give fluid, and what access to use to administer fluid will remain at the discretion of the treating team.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lactated Ringer — LR is a sterile, nonpyrogenic "balanced" solution used for fluid and electrolyte replenishment via intravenous or intraosseous administration. Each 100 mL of LR contains 600 mg sodium chloride (NaCl), 310 mg of sodium lactate (C3H5NaO3), 30 mg of potassium chloride (KCl), and 20 mg of calcium chloride (CaCl2 · 2H20) with an approximate potential of hydrogen (pH) of 6.5 (6.0 to 7.5).
  Other Names: LR
  Arms: Balanced fluids (BF)
Drug: Normal Saline — Normal saline solution is an "unbalanced" crystalloid solution containing 154 mEq/L of sodium and 154 milliequivalent (mEq/L) of chloride.
  Other Names: 0.9% Saline; NS
  Arms: 0.9% "Normal" Saline Fluid (NS)
Drug: Plasma-lyte — PL is a sterile, nonpyrogenic isotonic solution in a single dose container for intravenous administration. Each 100 mL contains 526 mg of Sodium Chloride, USP (NaCl); 502 mg of Sodium Gluconate (C6H11NaO7); 368 mg of Sodium Acetate Trihydrate, USP (C2H3NaO2•3H2O); 37 mg of Potassium Chloride, USP (KCl); and 30 mg of Magnesium Chloride, USP (MgCl2•6H2O). It contains no antimicrobial agents. The pH is adjusted with sodium hydroxide. The pH is 7.4 (6.5 to 8.0).
  Other Names: PL
  Arms: Balanced fluids (BF)

SUMMARY:
The objectives of this multicenter pragmatic clinical trial are to compare the effectiveness and relative safety of balanced fluid resuscitation versus 0.9% "normal" saline in children with septic shock, including whether balanced fluid resuscitation can reduce progression of kidney injury.

DETAILED DESCRIPTION:
Approximately 5,000 children die from septic shock each year in the United States (US); thousands more die worldwide. Most children admitted with sepsis receive initial resuscitation in an emergency department (ED), where septic shock remains one of the most critical of illnesses treated by ED clinicians. Sepsis is also the most expensive hospital condition in the US, and the most common cause of pediatric multiple organ dysfunction syndrome (MODS). While all crystalloid fluids help to reverse shock, the most effective and safest type of crystalloid fluid resuscitation is unknown.

Crystalloid fluids can be categorized as non-buffered (most commonly 0.9% normal saline [NS]) or buffered/balanced fluids (BF). In the US, the most common BF is lactated Ringer's (LR), but other example include PlasmaLyte. NS and BF are inexpensive, stable at room temperature, and nearly universally available with identical storage volumes and dosing strategies. Notably, both are also of proven clinical benefit in septic shock and have extensive clinical experience for use in fluid resuscitation of critically ill patients. However, despite data suggesting that BF resuscitation may have superior efficacy and safety, NS remains the most commonly used fluid largely based on historical precedent.

To definitively test the comparative effectiveness of NS and BF, a well-powered randomized controlled trial (RCT) is necessary. A large pragmatic randomized trial embedded within everyday clinical practice provides a cost-efficient and generalizable approach to inform clinicians about best comparative effectiveness of common therapies. Data from a prior single-center feasibility study demonstrated that a pragmatic randomized clinical trial of NS versus BF for children with septic shock presenting to an emergency department is feasible and can be successfully carried out by embedding simple study procedures within routine clinical practice. This multi-center study that will now test for differential clinical effects, as part of a definitive comparative effectiveness trial, of NS versus BF for crystalloid resuscitation of pediatric septic shock.

This multicenter phase trial will include enrollment and study procedures across 30+ US and international sites to compare the effectiveness and relative safety of NS versus BF (LR and PlasmaLyte) for crystalloid resuscitation of children with septic shock. The primary endpoint is major adverse kidney events within 30 days along with other secondary clinical, safety, and kidney biomarker endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age >2 months to <18 years
2. Clinician concern for septic shock, operationalized as:

   1. a "positive" ED sepsis alert confirmed by a physician OR
   2. physician decision to treat for septic shock OR
   3. a physician diagnosis of septic shock requiring parenteral antibiotics and fluid resuscitation
3. Administration of at least one IV/Intraosseous (IO) fluid bolus for resuscitation and additional fluid deemed likely to be necessary to treat poor perfusion, or clinician judgment that >1 fluid bolus is highly likely to be required. Poor perfusion is defined as physician's judgement of hypotension or abnormal (either "flash" or "prolonged") capillary refill.
4. Receipt of ≤40 mL/kg IV/IO total crystalloid fluid prior to randomization
5. Parental/guardian permission (informed consent) if time permits; otherwise, Exception from informed consent (EFIC) criteria met

Exclusion Criteria:

1. Treating physician judges that patient's condition deems it unsafe to administer either NS or BF (since patients will be equally likely to receive NS or BF at time of study enrollment), including:

   1. Clinical suspicion for impending brain herniation
   2. Known hyperkalemia, defined as non-hemolyzed whole blood or plasma/serum potassium > 6 mEq/L, based on data available at or before patient meets criteria for study enrollment
   3. Known hypercalcemia, defined as plasma/serum total calcium >12 mg/dL or whole blood ionized calcium >1.35 mmol/L, based on data available at or before patient meets criteria for study enrollment
   4. Known acute fulminant hepatic failure, defined as plasma/serum alanine aminotransferase (ALT) >10,000 U/L or total bilirubin >12.0 mg/dL, based on data available at or before patient meets criteria for study enrollment
   5. Known history of severe hepatic impairment, defined as cirrhosis, "liver failure", or awaiting transplant
   6. Known history of severe renal impairment, defined as peritoneal dialysis or hemodialysis
   7. Known metabolic/mitochondrial disorder, inborn error of metabolism, or primary mineralocorticoid deficiency as reported by participant, legally authorized representative (LAR) or accompanying caregiver, or as listed in the medical record
   8. Other concern for which the treating clinician deems it unsafe to administer either NS or LR
2. Known pregnancy determined by routine history disclosed by patient and/or accompanying acquaintance.
3. Known prisoner
4. Known allergy to a crystalloid fluid
5. Indication of declined consent to participate based on presence of an opt-out bracelet with appropriate messaging embossed into the bracelet, the presence of the patient's name on an opt-out list that will be kept up-to-date and checked prior to randomization, or verbal "opt-out" prior to enrollment.

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8800 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Major Adverse Kidney Events within 30 days (MAKE30) | Between randomization and 30 days post enrollment, discharge or death, whichever comes first.
  A composite of death, initiation of new inpatient renal replacement therapy (RRT), or persistent kidney dysfunction, at 30 days following study enrollment or hospital discharge, whichever comes first.

SECONDARY OUTCOMES:
Proportion of participants with persistent kidney dysfunction | Censored at 30 days
  Final creatinine greater than or equal to 200% of baseline and a minimum absolute increase of greater than or equal to 0.3 mg/dL
Proportion of participants with new inpatient renal replacement therapy | Censored at 30 days
  Treatment with any renal replacement therapy that was not a continuation of pre-hospital chronic therapy
Hospital-free days alive between randomization and day 27 | With 27 days of randomization
  Calendar days alive and out of the hospital between day of randomization and study day 27
Proportion of participants with all-cause hospital mortality | Hospital discharge-censored at 90 days
  Vital status at hospital discharge
Proportion of participants with all-cause mortality at 90 days | 90 days
  Vital status from medical chart and/or data from National Death Index
Proportion of participants with hyperlactatemia | Within 4 calendar days of randomization
  At least 1 venous or arterial blood lactate measurement >4mmol/L
Proportion of participants with hyperkalemia | Within 4 calendar days of randomization
  At least 1 venous or arterial blood potassium measurement >6 milliequivalents/Liter (mEq/L) (without hemolysis)
Proportion of participants with hypercalcemia | Within 4 calendar days of randomization
  At least 1 venous or arterial blood ionized calcium measurement of >1.35 mEq/L or total calcium >12 mEq/L
Proportion of participants with hypernatremia | Within 4 calendar days of randomization
  At least 1 venous, arterial or capillary blood sodium measurement of >155 mEq/L
Proportion of participants with hyponatremia | Within 4 calendar days of randomization
  At least 1 venous, arterial or capillary blood sodium measurement of <128 mEq/L
Proportion of participants with hyperchloremia | Within 4 calendar days of randomization
  At least 1 venous, arterial or capillary blood chloride measurement of >110 mEq/L
Proportion of participants with catheter thrombosis | Within 4 calendar days of randomization
  Catheter thrombosis in participants given Ceftriaxone and BF? (not LR?)
Proportion of participants with brain herniation | Within 4 calendar days of randomization
  Treatment with hyperosmolar therapy (as long as a clinical diagnosis of brain herniation is not disproven by radiographic studies)
Proportion of participants with thromboembolism | Within 7 calendar days of randomization
  Therapy for thromboembolism

OTHER OUTCOMES:
Kidney biomarkers measured from blood and urine samples | Day 2 and Day 27, prior to anticipated discharge or death, whichever comes first.
  Urine neutrophil gelatinase-associated lipocalin (NGAL), urine NGAL/Ucr ratio, Kidney injury molecule (KIM-1), KIM-1/ Ucr ratio, Liver-type fatty acid binding protein (L-FBP), L-FBP/ Ucr ratio, Interleukin (IL-18), IL-18/ Ucr ratio, and plasma cystatin C measured on study day 2 and on day 27 (or prior to anticipated discharge or death, whichever comes first).

CONTACTS AND LOCATIONS:
Overall Officials: Fran Balamuth, MD PhD MSCE, Principal Investigator — Attending Physician, Emergency Department
Locations (22):
- United States (22):
  - UC Davis: University of California, Davis, Davis, California
  - CHLA: Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Colorado: University of Colorado, Denver, Colorado
  - Children's Hospital of Atlanta, Emory, Georgia
  - Lurie Children's: Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Columbia: New York-Presbyterian Hospital, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Dallas Children's: Children's Medical Center Dallas/UT southwestern, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's: University of Utah, Salt Lake City, Utah
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - Children's National Medical Center, Columbia, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Milwaukee (MCW): Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Per NIH policy, the PRoMPT BOLUS investigators will provide a de-identified dataset and documentation necessary to utilize the study data (dictionary, calculated variables, and standard operating procedures) to the NIH no later than 3 years after the final 90-day assessment or 2 years after the primary paper has been published, whichever comes first. The investigators will submit this dataset to the National Institute of Child Health and Human Development (NICHD) data repository, Data and Specimen Hub (DASH). In addition, final datasets and statistical analyses will be archived.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No later than 3 years after the final 90-day assessment or 2 years after the primary paper has been published, whichever comes first.
Access Criteria: Anyone can access NICHD DASH, which is a public website with free access to the scientific research community. All users may browse and view information about studies and data archived in NICHD DASH. Users who are interested in submitting or requesting study data must register for a free account.

REFERENCES:
- [Background] Balamuth F, Kittick M, McBride P, Woodford AL, Vestal N, Casper TC, Metheney M, Smith K, Atkin NJ, Baren JM, Dean JM, Kuppermann N, Weiss SL. Pragmatic Pediatric Trial of Balanced Versus Normal Saline Fluid in Sepsis: The PRoMPT BOLUS Randomized Controlled Trial Pilot Feasibility Study. Acad Emerg Med. 2019 Dec;26(12):1346-1356. doi: 10.1111/acem.13815. Epub 2019 Jul 18. PMID 31183919
- [Derived] Weiss SL, Balamuth F, Long E, Thompson GC, Hayes KL, Katcoff H, Cook M, Tsemberis E, Hickey CP, Williams A, Williamson-Urquhart S, Borland ML, Dalziel SR, Gelbart B, Freedman SB, Babl FE, Huang J, Kuppermann N; Pragmatic Pediatric Trial of Balanced Versus Normal Saline Fluid in Sepsis (PRoMPT BOLUS) Investigators of the PECARN, PERC, and PREDICT Networks. PRagMatic Pediatric Trial of Balanced vs nOrmaL Saline FlUid in Sepsis: study protocol for the PRoMPT BOLUS randomized interventional trial. Trials. 2021 Nov 6;22(1):776. doi: 10.1186/s13063-021-05717-4. PMID 34742327
- See also: PRoMPT BOLUS website — https://promptbolus.research.chop.edu/